CLINICAL TRIAL: NCT01669148
Title: Breast Cancer Detection: Comparison of Breast Tomosynthesis and Conventional Mammography
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Massachusetts General Hospital (Other)
Collaborators: Hologic, Inc. (Industry)
Responsible Party: Principal Investigator, Thomas J. Brady, M.D., Vice Chairman, Radiology Research, Massachusetts General Hospital
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: 2007p-001197
Record Dates: First submitted 2010-04-30; First posted 2012-08-20 (Estimated); Results first posted 2017-06-14 (Actual); Last update posted 2017-06-14 (Actual); Status verified 2017-01

CONDITIONS: Breast Cancer
Keywords: breast cancer; imaging
MeSH Terms: conditions — Breast Neoplasms | interventions — Mammography

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Conventional + Tomosynthesis (Active Comparator): conventional (2D) imaging plus tomosynthesis (3D) imaging first then tomosynthesis alone 1 month later.
  Interventions: Device: Tomosynthesis; Device: Conventional
- Tomosynthesis alone (Active Comparator): tomosynthesis (3D) imaging alone first then conventional (2D) imaging plus tomosyntheis 1 month later.
  Interventions: Device: Tomosynthesis

INTERVENTIONS:
Device: Tomosynthesis — The mean glandular radiation dose for each image will be approximately 145 millirads (mrad) for a standard size breast (4.2 cm compressed breast thickness).
Device: Conventional — conventional (2D) imaging (standard mammography)
  Arms: Conventional + Tomosynthesis

SUMMARY:
The primary hypothesis to be tested is:

The detection of breast cancer will be increased with tomosynthesis (3D) imaging

DETAILED DESCRIPTION:
The purpose of this study is to determine if: 1 the detection of breast cancer will be increased with conventional (2D) imaging plus tomosynthesis (3D) imaging, or 2. if the the detection of breast cancer will be increased with tomosynthesis (3D) imaging alone.

ELIGIBILITY:
Inclusion Criteria:

* Female
* Any ethnic origin
* No contraindication for routine bilateral mammography

Exclusion Criteria:

Potential subjects with any of the following will not be enrolled in the study:

* Any contraindications to mammographic screening, including, but not limited to:
* Significant existing breast trauma
* Under the age of 30 at the time of consent
* Breast Implants
* Prior Surgeries

  * Unable to understand and execute written informed consent
  * Pregnant
  * Lactating

Min Age: 35 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 496 (Actual)
Dates: Start 2007-11; Primary Completion 2011-06 (Actual); Study Completion 2012-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Elizabeth A Rafferty, MD, Principal Investigator — Massachusetts General Hospital
Locations (1):
- MGH, Boston, Massachusetts, United States

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: 496 enrolled and 426 completed study, but no information available to distinguish study arms:
  1. Conventional+Tomosynthesis First Then Tomo alone 1 mo. Later (number of participants enrolled in arm is unknown).
  2. Tomosynthesis alone First Then Conventional+Tomo 1 mo. Later (number of participants enrolled in arm is unknown).
Groups:
- All Study Participants: All participants enrolled in study
Period: Overall Study
Arm/Group | All Study Participants
Started | 496
Completed | 426
Not Completed | 70

BASELINE CHARACTERISTICS:
Population: 496 participants enrolled overall, but no information available to distinguish study arms:
  1. Conventional+Tomosynthesis First Then Tomo alone 1 mo. Later (number of participants enrolled in arm is unknown).
  2. Tomosynthesis alone First Then Conventional+Tomo 1 mo. Later (number of participants enrolled in arm is unknown).
Groups:
- All Study Participants: All study participants in both arms. 496 enrolled and 426 completed study, but no information available to distinguish study arms.
Arm/Group | All Study Participants
Number analyzed (Participants) | 496
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 427
  >=65 years | 69
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 496
  Male | 0
Region of Enrollment [Number; unit: participants]
  United States | 248

OUTCOME MEASURES:

1. Primary Outcome: Detection of Breast Cancer (Sensitivity)
Description: Sensitivity is the number of true positives (TP) divided by the sum of TP and false negatives (FN):
  Sensitivity = TP / (TP+FN)
Time Frame: up to two years follow up for development of breast cancer
Population: PI left institution in 2012; Data remaining did not include outcome measure and adverse event data. Institution contacted PI on numerous occasions. PI also does not have data.
Groups:
- Conventional + Tomosynthesis First Then Tomo Alone 1 mo. Later; Tomosynthesis Alone First Then Conventional+Tomo 1 mo. Later: Tomosynthesis: The mean glandular radiation dose for each image will be approximately 145 millirads (mrad) for a standard size breast (4.2 cm compressed breast thickness).
  Conventional: conventional (2D) imaging (standard mammography)
Arm/Group | Conventional + Tomosynthesis First Then Tomo Alone 1 mo. Later | Tomosynthesis Alone First Then Conventional+Tomo 1 mo. Later
Number analyzed (Participants) | 0 | 0

ADVERSE EVENTS:
Description: PI left institution in 2012; Data remaining did not include outcome measure and adverse event data. Institution contacted PI on numerous occasions. PI also does not have data.
  496 participants enrolled overall, but no information available to distinguish study arms:
  1. Conventional+Tomosynthesis First Then Tomo alone 1 mo. Later (number enrolled in arm is unknown).
  2. Tomosynthesis alone First Then Conventional+Tomo 1 mo. Later (number enrolled in arm is unknown).
Groups:
- All Study Participants: All participants enrolled in the study
Arm/Group | All Study Participants
Serious Adverse Events (participants affected / at risk) | 0/0
Other Adverse Events (participants affected / at risk) | 0/0

LIMITATIONS AND CAVEATS:
PI left institution in 2012; Data remaining did not include outcome measure and adverse event data. Institution contacted PI on numerous occasions. PI also does not have data.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes